CLINICAL TRIAL: NCT03272984
Title: Enhanced Recovery After Surgery Programs for Patients Received Neoadjuvant Chemotherapy With Locally Advanced Gastric Cancer: a Randomized Controlled Clinical Trial
Brief Title: ERAS for Patients Received Neoadjuvant Chemotherapy
Acronym: ERASNAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JIANG Zhi-Wei (Other)
Responsible Party: Sponsor-Investigator, JIANG Zhi-Wei, Vice director of Research Institute of General Surgery, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8150041701
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a parallel, open-label randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Experimental): Patients will undergo the ERAS programs.
  Interventions: Procedure: ERAS group
- SC group (Other): Patients will undergo the SC group.
  Interventions: Procedure: SC group

INTERVENTIONS:
Procedure: ERAS group — ERAS is the name of a procedure. Patients in this group need receive the ERAS procedure instead of one drug.
  Arms: ERAS group
Procedure: SC group — Patients were managed in accordance with SC programs during the perioperative period. SC programs were used daily in our center and were still routinely used in most of the other hospitals in China.
  Arms: SC group

SUMMARY:
Patients received neoadjuvant chemotherapy with locally advanced gastric caner undergo the enhanced recovery after surgery (ERAS) programs or the standard cares (SC) programs.

DETAILED DESCRIPTION:
Before, most trials about the ERAS for radical gastrectomy demonstrated ERAS programs accelerate the postoperative rehabilitation of gastric cancer patients without increasing postoperative complications. However, in most trials, patients who received neoadjuvant chemotherapy were excluded. The investigators designed this trial for patients received neoadjuvant chemotherapy. In this trial, patients received neoadjuvant chemotherapy with locally advanced gastric caner undergo the ERAS programs or the SC programs. Finally, the investigators evaluated whether patients who receive neoadjuvant chemotherapy can be enrolled into the ERAS programs for locally advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients received neoadjuvant chemotherapy with locally advanced gastric cancer.
2. Age older than 18 and younger than 75 years.
3. American Society of Anesthesiologists (ASA) class: I-III.
4. Participants can describe the symptom objectively and cooperate actively.
5. Written informed consent.

Exclusion Criteria:

1. Patients allergic to oxaliplatin, tegafur gimerac etc.
2. Patients with ischemic heart disease, cerebrovascular disease and peripheral vascular disease, or cardiac function > II (NYHA)
3. Patients with complications (bleeding, perforation and obstruction) caused by gastric cancer.
4. Patients with severe liver and renal dysfunction (Child - Pugh ≥ 10; Cr < 25 ml/min).
5. Patients who require simultaneous surgery for other diseases.
6. Patients who received upper abdominal surgery previously.
7. Pregnant or breast-feeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Postoperative length of stay | 1 month
  Postoperative length of stay

SECONDARY OUTCOMES:
Postoperative complications | 2 months
  Postoperative complications
The time to first flatus | 1 week
  Bowel recovery
Time to semi-liquid diet | 2 week
  Bowel recovery

CONTACTS AND LOCATIONS:
Overall Officials: Zhiwei JIANG, MD, Principal Investigator — Jinling Hospital, Medical School of Nanjing University; Jian ZHAO, MD, Study Director — Jinling Hospital, Medical School of Nanjing University
Locations (1):
- Jinling Hospital, Medical School of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
The results and IPD will be considered to share in published articles.